CLINICAL TRIAL: NCT03591068
Title: A 24-Week Open-Label Study Evaluating the Efficacy and Safety of OPN-375 186 μg Twice a Day (BID) in Adults With Bilateral Nasal Polyps Using Nasoendoscopic Video
Brief Title: Efficacy & Safety of OPN-375 Adults With Bilateral Nasal Polyps Using Nasoendoscopic Video
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-FLU-NP-3104
Record Dates: First submitted 2018-06-11; First posted 2018-07-18 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Nasal Polyposis
MeSH Terms: conditions — Nasal Polyps | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OPN-375 186 mcg BID (Experimental)
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — OPN-375 186 μg BID, Delivered via exhalation delivery system

SUMMARY:
This is a 24-week, open-label, multi-center study designed to assess the efficacy and safety of OPN-375 186 μg twice a day in subjects with nasal polyps using Nasoendoscopic video. The total planned number of subjects is approximately 10, with each subject receiving OPN-375 186 μg twice a day.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of OPN-375 186 μg twice a day in adults with Bilateral Nasal Polyps using Nasoendoscopic video. The secondary objectives of this study are to evaluate the safety of OPN-375 via adverse event reports, vital signs, and nasal examination. In addition, to measure any change in subject symptoms and functioning from Baseline to 12 and 24 weeks during the study, using the Sinonasal Outcome Test -22 (SNOT-22), Patient's Global Impression of Change (PGIC), and measurement of nasal polyps by independent, blinded reader, and any changes throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 years and older at Visit 1 (Baseline/Day1)
2. Women of child bearing potential must be abstinent, or if sexually active,

   1. be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   2. be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   3. be postmenopausal (amenorrhea for at least 1 year).
3. Women of child-bearing potential must have a negative urine pregnancy test at Visit 1 (Day 1/Baseline)
4. Must have bilateral nasal polyposis with a grade of 2 or 3 in at least one side of the nasal cavity as determined by a nasal polyp grading scale score measured by nasoendoscopy at Visit 1 (Day 1/Baseline)
5. Must have a SNOT-22 score of ≥20 at Visit 1(Baseline/Day 1)
6. Must have been on an adequate dose of an intranasal corticosteroid (e.g. fluticasone propionate, fluticasone furoate, mometasone, triamcinolone, ciclosenide, budesonide, budesonide respules, beclomethasone) for at least 1 month, in the previous 3 months prior to Visit 1 (Day 1/Baseline)
7. Subjects with comorbid asthma or chronic obstructive pulmonary disease (COPD) must be stable with no exacerbations (e.g., no emergency room visits, hospitalization, or oral or parenteral steroid use) within the 3 months before the screening visit. Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent) for at least 3 months before screening with plans to continue use throughout the study
8. Must be able to cease treatment with oral steroids, intranasal steroids, inhaled corticosteroids (except permitted doses listed above for asthma and COPD) at Visit 1 (Day 1/Baseline)
9. Must demonstrate correct use of the demo EDS
10. Ability to read and speak English
11. Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Inability to have each nasal cavity examined for any reason, including nasal septum deviation
3. Have used XHANCE™ (fluticasone propionate) nasal spray within the past 2 months
4. Nasal septum perforation
5. Has had more than 1 episode of epistaxis with frank bleeding in the month before Visit 1 (Day 1/Baseline)
6. Have evidence of significant mucosal injury or ulceration (e.g. exposed cartilage) on Visit 1 (Day 1/Baseline) nasal examination/nasoendoscopy
7. History of sinus or nasal surgery within 3 months before Visit 1 (Day 1/Baseline). If >3 months subject should be fully recovered from surgery
8. Current, ongoing rhinitis medicamentosa (rebound rhinitis)
9. Have significant oral structural abnormalities, e.g., a cleft palate
10. Diagnosis of cystic fibrosis
11. History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
12. Purulent nasal infection, acute sinusitis, or upper respiratory tract infection within 2 weeks before Visit 1 (Day 1/Baseline). Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution
13. Planned sinonasal surgery during the period of the study
14. Allergy, hypersensitivity, or contraindication to corticosteroids, steroids, or to any excipients in OPN-375
15. Exposure to any glucocorticoid treatment with potential for systemic effects (e.g., oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before Visit 1 (Day 1/Baseline); except as noted in inclusion criteria for subjects with comorbid asthma or COPD
16. Have nasal candidiasis at Visit 1 (Day 1/Baseline)
17. History or current diagnosis of any form of glaucoma, ocular hypertension, or intraocular pressure elevation on any form of steroid therapy
18. History or current diagnosis of the presence (in either eye) of a sub-capsular cataract
19. Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
20. Recent (within 1 year of Visit 1 (Day 1/Baseline)) history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
21. Have participated in an investigational drug clinical trial within 30 days of Visit 1 (Day 1/Baseline)
22. Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carothers, Study Director — Optinose US Inc.; John Messina, Study Chair — Optinose US Inc.
Locations (2):
- United States (2):
  - University of Colorado SOM, Department of Otolaryngology, Aurora, Colorado
  - University of Texas Health Science Center at Houston, McGovern Medical School, Dept. of Otolaryngology, Head and Neck Surgery, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPN-375 186 mcg BID
Started | 11
Completed | 9
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Total Polyp Grading Score (sum of scores from both nasal cavities) [Mean (Full Range); unit: units on a scale] — Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
  units on a scale | 3.1 [2 to 6]
Sinonasal Outcome Test 22 (SNOT-22) Total Score [Mean (Full Range); unit: units on a scale] — SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as can be
  units on a scale | 48.8 [26 to 74]
Sniffin' Sticks n-butanol tests [Mean (Standard Deviation); unit: units on a scale] — Consists of 3 different subtests: Threshold, Discrimination and Identification. Threshold test is used to analyze the olfactory threshold. Discrimination test requires the patient to differentiate smells. Identification test requires the patient to identify everyday smells through a card with various choices. Result of this test is expressed as sum of results of 3 subtests (TDI score). A score of > 30 rates as normal, a score of <=30 indicates hyposmia and a score of <=15 point to functional anosmia in form of complete loss of the sense of smell or an extremely weakened smell ability.
  units on a scale | 11.8 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Visit 1 at End of Study in Bilateral Nasal Polyp Grade Using Endoscopic Video
Description: : Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy. 0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
units on a scale | -0.7 (0.9)

2. Secondary Outcome: Assessment for Safety by Recording Adverse Events and Adverse Events of Special Interests
Time Frame: 24 Weeks, up to 30 days after last dose
Population: No TEAE was experienced by more than a single subject
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants
  Asthma | 1
  Back pain | 1
  Dizziness | 1
  Dyspnoea | 1
  Fungal skin infection | 1
  Hypotension | 1
  Influenza | 1
  Lacrimation increased | 1
  Nasal discharge discolouration | 1
  Sinusitis | 1
  Tension headache | 1
  Upper respiratory tract infection | 1
  Vasomotor rhinitis | 1

3. Secondary Outcome: Assessment for Safety Through Nasal Examination
Description: Assessed in nasal examination worksheet which includes recording the presence of any epistaxis, septal erosion/perforation, ulceration/erosion of area other than septum. If present, the nostril location is also recorded, along with severity, and if there is any relation to an injury or trauma
Time Frame: 24 Weeks, up to 30 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants
  Epistaxis | 1
  Septal erosion/perforation | 0
  Ulceration/erosion | 0

4. Secondary Outcome: Assessment for Safety From Recording Vital Sign - Blood Pressure
Description: Includes systolic and diastolic blood pressure measurements in millimeter of mercury (mmHg)
Time Frame: Baseline, Week 12, Week 24
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- OPN-375 186 mcg BID - Systolic BP; OPN-375 186 mcg BID - Diastolic BP: Fluticasone Propionate: OPN-375 186 μg BID, Delivered via exhalation delivery system
Arm/Group | OPN-375 186 mcg BID - Systolic BP | OPN-375 186 mcg BID - Diastolic BP
Number analyzed (Participants) | 11 | 11
mmHg
  Baseline | 130.1 (14.3) | 83.3 (9.3)
  Week 12 | 127.4 (19.6) | 82.0 (12.9)
  Week 24 | 131.9 (18.8) | 81.4 (8.7)

5. Secondary Outcome: Assessment for Safety From Recording Vital Sign - Pulse
Description: measure pulse in beats per minute (bpm)
Time Frame: Baseline, Week 12, Week 24
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
bpm
  Baseline | 71.5 (7.1)
  Week 12 | 73.5 (9.1)
  Week 24 | 76.4 (7.4)

6. Secondary Outcome: Assessment for Safety From the Collection of Information for Concomitant Medications Usage
Time Frame: 24 Weeks, up to 30 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants
  ACE Inhibitor | 1
  Angiotensin II Receptor Antagonist | 1
  Antianginal | 1
  Anticoagulant | 1
  Antihistamine | 4
  Antifungal Cream | 1
  Ascorbic Acid | 1
  Beta Blocking Agent, selective | 2
  Beta2 Adrenergic Agonist | 6
  Biguanide | 1
  Calcium Channel Blocker | 1
  CNS Muscle Relaxant | 1
  Diuretic | 2
  Electolytes | 1
  HMG CoA Reductase Inhibitors | 1
  Inhaled Corticosteroid | 2
  Inhaled Corticosteroid/Long-acting beta-agonist | 6
  Leukotriene Receptor Antagonists | 3
  Multivitamin | 2
  Nitrate | 1
  Non-steroidal anti-inflammatory drug | 3
  Nuclear factor erythroid-2-related factor | 1
  Selective serotonin reuptake inhibitor | 1
  Synthetic nucleoside analogue | 1
  Other analgesics | 1
  Other antiinflammatorys | 1
  Topical antibiotics | 2
  Proton pump inhibitors | 1
  Testosterone | 1
  Thyroid Hormone | 2

7. Secondary Outcome: Total Polyp Grading Score (Sum of Scores From Both Nasal Cavities)
Description: Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy. 0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
Time Frame: Week 24
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
units on a scale | 2.4 [2 to 4]

8. Secondary Outcome: Number of Subjects With a Change of Greater Than or Equal to 1 Point in Bilateral Polyp Grade
Description: as for outcome 7
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants | 5

9. Secondary Outcome: Number of Subjects With a Polyp Grade of 0 on at Least One Side of the Nose at Each Visit
Description: as for outcome 7
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants | 1

10. Secondary Outcome: Sinonasal Outcome Test 22 (SNOT-22) Total Score
Description: SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as can be
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
units on a scale | 27.8 (16.1)

11. Secondary Outcome: Sniffin' Sticks N-butanol Test
Description: The Sniffin' Sticks n-butanol (Extended test) are used to investigate human olfactory performance by use of odor pens. the Extended Test consists of 3 different subtests: Threshold, Discrimination and Identification. the Threshold test is used to ascertain the patient's olfactory threshold. the Discrimination test requires the patient to differentiate smells. The Identification test requires the patient to identify everyday smells by means of a card with different choices. The result of this test is expressed as the sum of the results of the 3 subtests, the so called TDI score (threshold, discrimination, identification). A score of more than 30 rates as normal, a score of 30 or less indicates hyposmia and a score of 15 and below point to functional anosmia in form of complete loss of the sense of smell or an extremely weakened smell ability.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
units on a scale | 16.5 (6.9)

12. Secondary Outcome: Number of Participants With a PGIC Score of Minimally/Much/Very Much Improved
Description: The Patient Global Impression of Change (PGIC), is a questionnaire where the patient rates the change in their symptoms. Score range is from 1 (very much improved) to 7 (very much worse)
Time Frame: Week 24
Population: Number of participants who responded that they had some degree of improvement in their symptoms (minimally/much/very much improved)
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 mcg BID
Number analyzed (Participants) | 11
Participants | 9

ADVERSE EVENTS:
Time Frame: 24 weeks, and up to 30 days after the last dose
Arm/Group | OPN-375 186 mcg BID
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPN-375 186 mcg BID (N=11)
Dyspnea (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Fungal Skin Infection (Infections and infestations) | 1
Hypotension (Cardiac disorders) | 1
Influenza (Infections and infestations) | 1
Lacrimation Increased (Eye disorders) | 1
Nasal Discharge Discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis (Infections and infestations) | 1
Tension Headache (Nervous system disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Vasomotor Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement is described in CTA between sponsor and PI

DOCUMENTS (2):
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03591068/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT03591068/Prot_SAP_002.pdf